CLINICAL TRIAL: NCT00310063
Title: Acupressure for the Prevention of Chemotherapy-Associated Nausea and Vomiting in Children
Brief Title: Acupressure in Preventing Nausea and Vomiting in Young Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000466312; CCCWFU-02104; CCCWFU-BG05-101
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Nausea and Vomiting; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified childhood solid tumor, protocol specific
MeSH Terms: conditions — Nausea; Vomiting | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Sea Band elastic acupressure wristband
  Interventions: Procedure: acupressure therapy
- Arm II (Sham Comparator): Sham wristband
  Interventions: Procedure: sham intervention

INTERVENTIONS:
Procedure: acupressure therapy — Acupressure wristband
  Arms: Arm I
Procedure: sham intervention — Sham wristband
  Arms: Arm II

SUMMARY:
RATIONALE: Using acupressure wrist bands to press and stimulate nerves at an acupressure point on the inside of the wrist may help control nausea and vomiting caused by chemotherapy.

PURPOSE: This randomized clinical trial is studying how well acupressure works in preventing nausea and vomiting in young cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of implementing an acupressure therapy for the prevention of chemotherapy-associated nausea in children with cancer.
* Test the hypothesis that acupressure bands will prevent chemotherapy-associated nausea and vomiting in children, when compared to placebo acupressure (wrist bands without acupressure).
* Develop a competitive grant application for a large, multi-institutional randomized controlled trial of the efficacy of acupressure in preventing chemotherapy-associated nausea in children.

OUTLINE: This is a prospective, randomized, placebo-controlled, crossover, pilot study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients wear Sea-Band elastic acupressure wristbands on each wrist beginning approximately 1 hour before beginning their first inpatient chemotherapy session and continuing for at least 24 hours after completing chemotherapy. Patients do not wear wristbands for their second chemotherapy session. Patients wear placebo wristbands on each wrist beginning approximately 1 hour before their third chemotherapy session and continuing for at least 24 hours after completing chemotherapy.
* Arm II: Patients wear placebo wristbands on each wrist beginning approximately 1 hour before their first chemotherapy session and continuing for at least 24 hours after completing chemotherapy. Patients do not wear wristbands for their second chemotherapy session. Patients wear Sea-Band acupressure wristbands on each wrist beginning approximately 1 hour before their third chemotherapy session and continuing for at least 24 hours after completing chemotherapy.

All patients also receive standard antiemetic therapy.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients must receive in-patient primary oncology care at least monthly at Brenner Children's Hospital

  * Patients may have any type of cancer
* Must be receiving at least 1 of the following chemotherapy agents as an inpatient:

  * An alkylating agent (e.g., cisplatin, cyclophosphamide, or ifosfamide)
  * An antitumor antibiotic (e.g., doxorubicin, daunomycin, dactinomycin, or mitoxantrone)
  * High-dose cytarabine

PATIENT CHARACTERISTICS:

* Patient's primary caregiver must speak English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 28 (Actual)
Dates: Start 2005-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
reduction of chemotherapy related nausea | 6 months
  assessment by questionaire of nausea during patient chemo

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Williams McLean, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Jones E, Isom S, Kemper KJ, McLean TW. Acupressure for chemotherapy-associated nausea and vomiting in children. J Soc Integr Oncol. 2008 Fall;6(4):141-5. PMID 19134445